CLINICAL TRIAL: NCT02361021
Title: Lung Aeration During WEANing From Mechanical Ventilation Determined by Electrical Impedance Tomography and Lung Ultrasound
Acronym: IWEAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Estaing (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0222
Record Dates: First submitted 2015-02-02; First posted 2015-02-11 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Critical Care; Weaning From Mechanical Ventilation; Electrical Impedance Tomography; End Expiratory Lung Volume; Lung Ultrasound Score
Keywords: Critical Care; Non invasive ventilation; Electrical impedance tomography; End expiratory lung volume; Lung ultrasound score

STUDY DESIGN:
Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: - Weaning from mechanical ventilation

SUMMARY:
Evaluation of lung aeration during weaning from mechanical ventilation determined by electrical impedance tomography and lung ultrasound

DETAILED DESCRIPTION:
Prospective clinical study in ICU with patients during weaning from mechanical ventilation comparing lung aeration determined by electrical impedance tomography and lung ultrasound.

Duration of weaning test is 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients during weaning test from mechanical ventilation
* Consent of patients or family
* Arterial line

Exclusion Criteria:

* Tracheotomized patients
* Dressings in the thoracic area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
End-expiratory lung volume (EELV) | at baseline
  End-expiratory lung volume (EELV) determined by electrical impedance tomography at baseline (start of the weaning test)
End-expiratory lung volume (EELV) | at hour 1
  - End-expiratory lung volume (EELV) determined by electrical impedance tomography at Hour 1 (end of the weaning test).

SECONDARY OUTCOMES:
Anterior, medio-anterior, medio-posterior and posterior EELV | at baseline (start of the weaning test)
Lung ultrasound score | at baseline (start of the weaning test)
Anterior, medio-anterior, medio-posterior and posterior EELV | at Hour 1 (end of the weaning test)..
Lung ultrasound score | at Hour 1 (end of the weaning test)..

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France